CLINICAL TRIAL: NCT07268196
Title: Impact of Liver Transplantation on Sexual Life and Function
Status: Recruiting | Type: Observational
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Other Study IDs: IEC/2024/110/MA03
Record Dates: First submitted 2025-11-22; First posted 2025-12-05 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Chronic Liver Disease and Cirrhosis
MeSH Terms: conditions — Fibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Chronic liver Disease: Chronic Liver disease patients undergoing elective liver transplantation
  Interventions: Other: No Treatment

INTERVENTIONS:
Other: No Treatment — This is an Observational Study

SUMMARY:
Liver Transplantation (LT) is a lifesaving intervention with around 90% of recipients currently surviving the first postoperative year and subsequent life expectancy now exceeding 20 years. After the post-operative recovery period, however, LT recipients become more and more confronted with the challenges of re-engagement with life after transplantation, a need to reach a new stability, reestablish function in everyday life, reconnect with valued roles, regain independence, and resume work Sexual function is a very important parameter in the evaluation of Quality of Life (QoL), as it has been shown that sexual dysfunction in transplant patients is associated with increased depression and decreased QoL. There are several studies in the relevant literature supporting the recovery of sexual function in patients after liver transplantation. It has been found that recovery was observed in erectile dysfunction in male patients 6 months after liver transplantation.

DETAILED DESCRIPTION:
Liver Transplantation (LT) is a lifesaving intervention with around 90% of recipients currently surviving the first postoperative year and subsequent life expectancy now exceeding 20 years. After the post-operative recovery period, however, LT recipients become more and more confronted with the challenges of re-engagement with life after transplantation, a need to reach a new stability, reestablish function in everyday life, reconnect with valued roles, regain independence, and resume work Sexual function is a very important parameter in the evaluation of Quality of Life (QoL), as it has been shown that sexual dysfunction in transplant patients is associated with increased depression and decreased QoL. There are several studies in the relevant literature supporting the recovery of sexual function in patients after liver transplantation. It has been found that recovery was observed in erectile dysfunction in male patients 6 months after LT

ELIGIBILITY:
Inclusion Criteria:

1. Married male Patients.
2. Decompensated Chronic Liver Disease awaiting elective liver transplantation.
3. Post Liver Transplant patients with stable graft function.

Exclusion Criteria:

1. Negative consent.
2. Patients with ongoing medical and surgical issues (biliary complications, graft complication etc.).
3. Acute on Chronic Liver Failure and Acute Liver Failure patients.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: Chronic Liver Disease patients awaiting elective transplantation and post liver transplant patients.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-12-07 (Actual); Primary Completion 2026-10-23 (Estimated); Study Completion 2026-10-23 (Estimated)

PRIMARY OUTCOMES:
Evaluation of sexual function by questionnaire method | pre transplant, 3,6,12 months
  Arizona Sexual Experience Scale (ASEX) scores for sexual dysfunction, ASEX scores are 5 point questionnaire with scores given for each question from 1-6. Total scores More than or equal to 19 indicate sexual dysfunction (higher the scores greater the sexual dysfunction).
Evaluation of erectile dysfunction using questionnaire method | pre transplant, 3,6,12 months
  International Index for Erectile Function - 5 (IIEF-5) scores for erectile dysfunction IIEF 5 scores are also a 5 point questionnaire with score ranging 0-6 for each question. Total scores less than 15 indicate mild to moderate erectile dusfunction and scores less than 11 indicate moderate erectile dysfunction (lower the scores higher the erectile dysfunction)

SECONDARY OUTCOMES:
Correlation between testosterone and Meld Na scores | pre transplant, 3,6,12 months
  Testosterone measured in ng/ml. Less than 2.84 ng/ml is considered as hypogonadism
Sarcopenia implication in recovery of sexual function. | pre transplant, 3,6,12 months
  Sarcopenia measured by third lumbar vertebra Skeletal muscle index. Values less than 52 indicates sarcopenia

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Dr. Viniyendra Pamecha, MS FEBS, Study Director — ILBS
Locations (1):
- ILBS, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided